CLINICAL TRIAL: NCT03950687
Title: A Multicenter, Randomized, Open Label, Active Comparator Parallel Controlled Phase 2 Clinical Study on Intravenous Administration of rESP Injection for the Treatment of Anemia in Chronic Renal Failure Patients With Hemodialysis.
Brief Title: Study of rESP Injection for the Treatment of Anemia in Chronic Renal Failure Patients With Hemodialysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-SSS06-HD-II-01
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Chronic Renal Failure With Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group A (Active Comparator): intravenous administration, maintaining the same dose and frequency administrated in the sceening period, for 32 weeks
  Interventions: Drug: Recombinant Human Erythropoiesis Injection (CHO cell)
- Experimental group B (Experimental): intravenous administration, 0.5μg/kg, once a week, for 32 weeks
  Interventions: Drug: Recombinant Erythropoiesis Stimulating Protein Injection(CHO cell)
- Experimental group C (Experimental): intravenous administration,
  1μg/kg, once every two weeks, for 32 weeks
  Interventions: Drug: Recombinant Erythropoiesis Stimulating Protein Injection(CHO cell)

INTERVENTIONS:
Drug: Recombinant Human Erythropoiesis Injection (CHO cell) — rHuEPO is a recombinant human erythropoietin with the same biological effects as natural erythropoietin
  Other Names: rHuEPO
  Arms: Control group A
Drug: Recombinant Erythropoiesis Stimulating Protein Injection(CHO cell) — rESP is a high glucose medium and long-acting recombinant protein products, containing 165 amino acids by adding 3 glycosylation sites
  Other Names: rESP
  Arms: Experimental group B; Experimental group C

SUMMARY:
A phase 2, randomized, open label, active comparator parallel controlled study to explore the dosage regiment of rESP, and evaluate its efficacy, safety and pharmacokinetic characteristics in the treatment of anemia in chronic renal failure patients with hemodialysis

DETAILED DESCRIPTION:
In this phase 2, open label, active comparator parallel controlled study, patients were randomly assigned to three study groups: one active comparator control group (rHu EPO, maintaining the same dose and frequency administrated in the sceening period ), and two experimental groups (0.5μg/kg ,once a week; 1.0μg/kg , once every two weeks). All the patients were administered intravenously for 32 weeks and were evaluated the efficacy, safety and pharmacokinetic characteristics. During the whole study period, dosage adjustment was not allowed in the first 4 weeks, while in the remaining trial period dosage adjustment was allowed once every two weeks if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic renal failure are undergoing maintenance hemodialysis for at least 3 months and at least 2 times a week;
2. 18 years old ≤ age ≤ 75 years old, gender is not limited;
3. Being treated with rHuEPO for at least 12 weeks, the average concentration of hemoglobin in the screening period is in the range of 100~120 g/L (including both ends), and the difference is less than 10g/L;
4. Evaluation of iron status within 4 weeks, transferrin saturation (TSAT) ≥ 20% and serum ferritin (SF) ≥ 200 μg / L;
5. Subjects agree to use reliable contraceptives by themselves and their spouses from the screening period to within 3 months after the end of the study;
6. Volunteer as a subject and sign an informed consent form.

Exclusion Criteria:

1. Patients who have received or plan to undergo a kidney transplant during the study period, or who plan to undergo other surgery during the study;
2. Except of renal anemia, there are other diseases that cause chronic anemia (such as sickle cell anemia, myelodysplastic syndrome, hematological malignancies, myeloma, hemolytic anemia, pure red blood cell aplastic anemia), blood systemic disease or coagulopathy;
3. There are acute or chronic blood loss within the past 3 months, such as gastrointestinal bleeding;
4. The following circumstances (including but not limited to), the investigators evaluated that it is not suitable for enrollment:

   * Kt/V<1.2 or URR<65%;
   * Abnormal liver function (the aspartate aminotransferase or alanine aminotransferase is greater than 3 times the upper limit of normal);
   * Patients who were positive for anti-HIV, anti-HCV, and Treponema pallidum antibodies;
5. Patiernts who was suffering from severe secondary hyperparathyroidism (sustained blood iPTH/PTH >1000 ng/L);
6. Patiernts who was suffering from malignant hypertension or poor control of blood pressure (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg);
7. Patients with previous thromboembolic disease (excluding luminal infarction), history of severe hematopoietic system, and high clotting tendency;
8. Patiernts with severe cardiovascular and cerebrovascular disease, severe or unstable coronary artery disease, heart failure (NYHA class III or IV), temporary vascular access, or myocardial infarction or stroke within 3 months;
9. Patients with malignant tumors (excluding non-melanoma skin cancer or excised carcinoma in situ);
10. Patients with a history of severe allergies (including drug allergies), allergic to erythropoietin, or allergic to any component of the test drug (such as human serum albumin);
11. The infection is being treated with systemic antibiotics;
12. Those who have received androgen therapy or who have received blood transfusion therapy within the past 8 weeks;
13. 5 months as a subject to participate in other new drug clinical trials or to the group when the withdrawal time is shorter than the five half-life of the test drug (whichever is the longest of the two);
14. All epilepsy or epilepsy history except of childhood febrile seizures, post-traumatic or abstinence single seizures;
15. Pregnant women and lactating women;
16. Alcohol, drug or drug addicts;
17. Other factors investigators believe that they may affect the efficacy judgment or is not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy index :hemoglobin concentration | 25th-32nd week
  the amount of change in mean Hb concentration compared with baseline Hb concentration during the evaluation period (25th-32nd week)

SECONDARY OUTCOMES:
Secondary efficacy index:maintenance rate | 25th-32nd week
  the proportion of subjects whose average Hb concentration remained within the target range during the evaluation period
Secondary efficacy index :proportion of subjects | for 32 weeks
  the proportion of subjects whose range of dose adjustments decreased or increased by 25% still did not reach 100-120 g/L (both ends)
Secondary efficacy index: proportion of times | 25th-32nd week
  the proportion of times the measured Hb concentration remains within the target range during the subject evaluation period
Secondary efficacy index : average weekly dose | 25th-32nd week
  the average weekly dose of the drug during the evaluation period (normalized by body weight)
Secondary efficacy index: EPO dose conversion coefficient of rESP | for 32 weeks
  the EPO dose conversion coefficient of rESP (the average weekly dose of rESP during the screening period) and the dose correlation
Secondary efficacy index : mean reticulocyte count | 25th-32nd week
  changes in mean values of reticulocyte compared to baseline values during the evaluation period.
Secondary efficacy index : mean red blood cell count | 25th-32nd week
  changes in mean values of red blood cell count compared to baseline values during the evaluation period
Safety indicator: adverse events | for 32 weeks
  the type, proportion and severity of adverse events
Safety indicator: number of dose adjustments | for 32 weeks
  the number of dose adjustments used by the subject during the treatment and evaluation period
Safety indicator: the ratio of subjects who are adjusted | for 32 weeks
  the ratio of subjects who are adjusted during the treatment and evaluation period
Safety indicator: incidence of erythropoietin (EPO) antibodies and anti-rESP antibodies | for 32 weeks
  incidence of erythropoietin (EPO) antibodies and anti-rESP antibodies
Maximum Plasma Concentration (Cmax) | for 32 weeks
  the Cmax of rESP in patients with long-term medication.
Area Under the Curve (AUC) | for 32 weeks
  the AUC of rESP in patients with long-term medication.

CONTACTS AND LOCATIONS:
Locations (1):
- The general hospital of the people's liberation army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No